CLINICAL TRIAL: NCT04693299
Title: Factors Related to a Persistent Inadequate Bowel Preparation After a Colonoscopy With Inadequate Colon Cleansing. An Observational Prospective Multicenter Study
Brief Title: Factors Related to a Persistent Inadequate Bowel Preparation for Colonoscopy
Acronym: REPREP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Lorenzo Fuccio, Principal Investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: REPREP
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Colonic Disease
MeSH Terms: conditions — Colonic Diseases | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: Inclusion criteria:
  Outpatient and hospitalized patients, adults, candidates for colonoscopy for any pathology, as part of the normal care process, with the need to repeat bowel preparation due to inadequate cleansing.
  Exclusion criteria:
  * Emergency regime
  * Inability to obtain consent
  * Refusal of the patient
  Interventions: Diagnostic Test: colonoscopy

INTERVENTIONS:
Diagnostic Test: colonoscopy — A colonoscopy scheduled within the normal pathway of care will be performed. No interventions will be performed.

SUMMARY:
Adequate bowel preparation for colonoscopy has an extremely relevant impact on diagnostic yield and procedural success. The guidelines recommend an adequate colon cleansing rate of at least 90% of procedures. It has been shown that patients with inadequate colon cleansing history have a high probability of not reaching an adequate bowel preparation again.

Surprisingly, no evidence-based recommendations are available regarding bowel preparation in the patient with inadequate colon cleansing history. Therefore, identifying the factors associated with repeated inadequacy of bowel cleansing is crucial in order to define the best preparation strategy in this subset of patients. The implications for patients and for healthcare system are many: improving the quality of bowel preparation would reduce the need to repeat colonoscopy and the risk of conducting unreliable examinations. Furthermore, it would reduce the costs for the healthcare system by avoiding to overload endoscopic units.

Inclusion criteria:

Outpatient and hospitalized patients, adults, candidates for colonoscopy for any pathology, as part of the normal care process, with the need to repeat bowel preparation due to inadequate cleansing.

Exclusion criteria:

* Emergency regime
* Inability to obtain consent
* Refusal of the patient

Primary end-point:

Identification of factors independently associated with repeated inadequate colon cleansing after inadequate bowel preparation at previous colonoscopy, and consequent development (and validation) of a predictive model.

The colon cleansing will be evaluated according to the Boston Bowel Preparation Scale (BBPS), which assigns a score from 0 (presence of solid stools) to 3 (excellent visualization of the colonic mucosa) for each of the three main segments of the colon, i.e. right colon, transverse colon and left-rectum colon. Colon cleansing will be judged inadequate in case of a total score <6 or a score <2 even in only one of the colic segments.

Secondary end-point:

• Assess the prevalence of repeated inadequate bowel cleansing in the patient with previous inadequate cleansing

ELIGIBILITY:
Inclusion Criteria:

* Outpatients or hospitalized patients
* adults
* candidates for colonoscopy for any pathology, in the normal pathway of care, with the need to repeat the bowel preparation due to inadequate colon cleansing.

Exclusion Criteria:

* Emergency regimen
* Inability to obtain consent
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient and hospitalized adult patients, candidates for colonoscopy for any pathology, in the normal pathway of care, with the need to repeat the bowel preparation due to inadequate colon cleansing.
Sampling Method: Non-Probability Sample
Enrollment: 407 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Identification of factors related to persistent inadequate colon cleansing at repeat colonoscopy due to inadequate colon cleansing. | Outcome will be assessed during colonoscopy.
  A logistic regression analysis will be run to identify such factors.

SECONDARY OUTCOMES:
Prevalence of persistent inadequate colon cleansing at repeat colonoscopy due to inadequate colon cleansing. | Outcome will be assessed during colonoscopy.
  The prevalence of inadequate colon cleansing at repeat colonoscopy will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Gastroenterologia ed Endoscopia Digestiva, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No